CLINICAL TRIAL: NCT00574613
Title: Phase II, Multicenter, Randomized, Double-blind, Intraindividually Placebo Controlled Clinical Trial, to Evaluate Efficacy and Safety of p144 Topical Administration for Skin Fibrosis in Patients With Systemic Sclerosis
Brief Title: Efficacy and Safety Study of p144 to Treat Skin Fibrosis in Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ISDIN (Industry)
Collaborators: Digna Biotech S.L. (Industry)
Responsible Party: ISDIN, ISDIN
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISD002-P144-07; 2007-002015-38
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Skin Fibrosis
Keywords: Skin fibrosis; systemic scleroderma; systemic sclerosis; P144; orphan drug; soluble collagen; durometer; skin fibrosis in systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: P144
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: P144 — Cream 0,3 ml once a day (3 months)
  Arms: 1
Drug: placebo — Cream 0,3 ml once a day (3 months)
  Arms: 2

SUMMARY:
Transforming growth factor-beta 1 (TGF-β1) is consistently over expressed in most fibrotic diseases and displays a variety of profibrotic effects in fibroblasts. Activation of TGF-β receptors induces the activation of several kinase signalling cascades leading to the phosphorylation of SMAD proteins as well as to the activation of SMAD-independent kinases that collectively activate ECM synthesis and fibroblast growth and differentiation into myofibroblasts. TGF-β1 is one of the main mediators in the fibrotic process, associated to both scarring and a long list of pathologies related to chronic inflammation and which affect all type of organs and tissues. An increase in TGF-β1 mRNA and protein levels has been described in these processes. Peptide 144 (P144) is the acetic salt of a 14mer peptide from human TGF-β1 type III receptor (betaglycan). P144 TGF-β1-inhibitor has been specifically designed to block the interaction between TGF-β1 and TGF-β1 type III receptor, thus blocking its biological effects. P144 has shown significant antifibrotic activity in mice receiving repeated subcutaneous injections of bleomycin, a widely accepted animal model of human scleroderma, and could contribute to the development. The purpose of this study is to asses the efficacy and safety of topical application of P144 in the treatment of skin fibrosis in patients with systemic sclerosis.

DETAILED DESCRIPTION:
Systemic sclerosis or scleroderma is a multisystemic disorder characterized by the excessive synthesis and deposition of extracellular matrix proteins that result in the fibrosis of skin and visceral organs (including gastrointestinal tract, lungs, heart and kidneys).

The pathogenesis of scleroderma is complex and still poorly understood, but major pathways involved in the development of the condition are microvascular and immunological abnormalities, as well as dysregulation of fibroblast activity. One of the key molecules involved in the pathogenesis of skin fibrosis is the TGF-β1; TGF-β1 is a cytokine directly responsible for fibroblasts proliferation and collagen and extracellular matrix overproduction.

The affected skin of patients with systemic sclerosis gradually becomes firm, thickened and eventually tightly bound to underlying subcutaneous tissue (indurative phase). It loses hair, oil, and sweat glands becoming dry and coarse. Changes begin distally in the extremities and advance proximally. Lesions develop over a period of time varying from months to a few years. In patients with limited scleroderma, only the skin of fingers, hands, face and lower arms and legs is affected. On the contrary, patients with the diffuse cutaneous disease, skin changes will become generalized, involving initially the extremities and followed by the face and trunk. Rapid progression of these changes over a 2 to 3 year period is usually associated with a greater risk of visceral disease. After several years of disease, the skin may soften and return to normal thickness or become thin and atrophic.

There is currently no approved specific treatment for skin fibrosis in systemic sclerosis neither in the European Union nor the United States of America. P144 belongs to a peptide family that is able to inhibit TGF-β1 in both in vitro and in vivo models characterized by excessive TGF-β1 function. Topical application of P144 exerts a preventive effect precluding the induction of skin fibrosis and the accumulation of collagen in these animals and also has shown its therapeutic properties reducing the skin fibrosis and soluble collagen content in mice with established fibrosis.

The EMEA and FDA have granted P144 the orphan drug status for the treatment of systemic sclerosis. In this study, the percentage of reduction in the soluble collagen content and skin hardness (durometer) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients male and female >18 < 65 years at time of consent.
* History of Systemic sclerosis (including diffuse scleroderma and limited scleroderma) for less than three years of evolution from the onset of cutaneous manifestations.
* Symmetric lesions in forearms. The extension of the selected symmetric lesions must be at least 15 cm2.
* Stable therapy for at least one month, except in the case of patients under treatment with putative disease modifying agents (immunosuppressants like cyclophosphamide, or azathioprine) that will need at least three months of stable therapy, without the expectation of treatment modifications during the trial period.
* Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* For female subjects with childbearing potential: use of a known highly effective method of birth control, defined as those which results in a low failure rate: i.e. less 1% per year, (contraceptive pills, intrauterine contraceptive device, implants, vasectomized partner or sexual abstinence), for at least three consecutive months prior to the study, during the study and one month after the end of the study.
* For male subjects with partners of child bearing potential: use of appropriate contraceptive methods (vasectomy, condoms or sexual abstinence), for at least the study period and one month after the end of the study.

Exclusion Criteria:

* Patients diagnosed of:

  * Systemic sclerosis sine scleroderma.
  * Localized scleroderma.
  * Eosinophilic fascitis, eosinophilia myalgia syndrome.
* Any other definable connective tissue disease, such as rheumatoid arthritis, systemic lupus erythematosus, polymyositis, or dermatomyositis.
* Clinically significant overlap condition.
* Significant existing internal organ damage (Kidney, Cardiovascular disease, Pulmonary disease, Gastrointestinal disease) as defined in "Guidelines for clinical trial in systemic sclerosis (scleroderma) " See appendix 1.
* History of skin cancer.
* Other skin diseases affecting the treatment area.
* Patients with substantial history of environmental exposure to tainted rapeseed oil, vinyl chloride, L- tryptophan, bleomycin, trichloroethylene, or silica.
* PUVA therapy within 1 month of study drug initiation.
* Concurrent interventional therapy that might independently influence outcome of trial, such as D-penicillamine, cyclosporine, methotrexate, interferon-α or photopheresis.
* Topical corticosteroids treatment affecting the selected area.
* Cosmetics over the treatment area.
* Pregnant or breast-feeding women.
* Reasonable expectation that the subject will not be able to satisfactorily complete the study:

  * History of or current psychiatric illness that would interfere with the subject's ability to comply with protocol requirements or give informed consent.
  * History of alcohol or drug abuse that would interfere with the subject's ability to comply with protocol requirements.
  * Receipt of any investigational drug within three months of screening visit.
  * Documented noncompliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The percentage of reduction in the soluble collagen content and skin hardness after three months relative to baseline. | Three months

SECONDARY OUTCOMES:
Changes in the histological and immunohistochemical analyses of P144 and placebo treated skin, in the expression levels of different molecular markers and changes from baseline in the skin elasticity quantified by Cutometer. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Matucci, MD, Study Chair; Thomas Krieg, MD, Principal Investigator; Ulf Müller-Ladner, MD, Principal Investigator; László Czirják, MD, Principal Investigator; Christopher Denton, MD, Principal Investigator; José Luis Pablos, MD, Principal Investigator
Locations (17):
- Germany (4):
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt, Frankfurt
  - Kerckhoff Klinik, Bad Nauheim, Hesse
  - Universität Köln, Cologne, Köln
  - Charité-Universitätsmedizin Berlin, Berlin, State of Berlin
- Magyarorszagi Irgalmasrend es Pécsi Tudomanyegyetem, Pécs, Pécs, Hungary
- Azienda Ospedaliera Universitaria Careggi., Florence, Italy
- Poland (5):
  - Centrum Miriada, Bialystok, Bialystok
  - Katedra i Klinika Chorób Wewnętrznych i Reumatologii, Katowice, Katowice
  - Katedra i Klinika Reumatologiczno, Poznan, Poznan
  - Gabinet Lekarski Internistyczno-Reumatologiczny, Wroclaw, Wroclaw
  - Klinika Ftizjopneumonologii SAM, Zabrze, Zabrze
- Spain (3):
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Pamplona
- United Kingdom (3):
  - Chapel Allerton Hospital, Leeds, Leeds
  - Royal Free Hospital, London, London
  - University Hospital Aintree, Liverpool

REFERENCES:
- [Background] Denton CP, Black CM. Scleroderma--clinical and pathological advances. Best Pract Res Clin Rheumatol. 2004 Jun;18(3):271-90. doi: 10.1016/j.berh.2004.03.001. PMID 15158741
- [Background] White B, Bauer EA, Goldsmith LA, Hochberg MC, Katz LM, Korn JH, Lachenbruch PA, LeRoy EC, Mitrane MP, Paulus HE, et al. Guidelines for clinical trials in systemic sclerosis (scleroderma). I. Disease-modifying interventions. The American College of Rheumatology Committee on Design and Outcomes in Clinical Trials in Systemic Sclerosis. Arthritis Rheum. 1995 Mar;38(3):351-60. doi: 10.1002/art.1780380309. PMID 7880189
- [Background] Querfeld C, Eckes B, Huerkamp C, Krieg T, Sollberg S. Expression of TGF-beta 1, -beta 2 and -beta 3 in localized and systemic scleroderma. J Dermatol Sci. 1999 Sep;21(1):13-22. doi: 10.1016/s0923-1811(99)00008-0. PMID 10468187
- [Background] Kissin EY, Schiller AM, Gelbard RB, Anderson JJ, Falanga V, Simms RW, Korn JH, Merkel PA. Durometry for the assessment of skin disease in systemic sclerosis. Arthritis Rheum. 2006 Aug 15;55(4):603-9. doi: 10.1002/art.22093. PMID 16874783
- See also: Asociación española de esclerodermia — http://www.esclerodermia.com/